CLINICAL TRIAL: NCT03339726
Title: Randomized, Double-blind, Placebo-Controlled Study of the Efficacy of Phenylephrine HCL Extended-Release 30 mg and Phenylephrine HCL Immediate-Release 12 mg Capsules in Subjects With Nasal Congestion Due to the Common Cold
Brief Title: Randomized, Double-blind, Placebo-Controlled, Efficacy Study of a New Formulation of Phenylephrine HCL in the Common Cold
Acronym: PIER
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: did not enroll enough subjects in the 2017/2018 cold season, so the study was terminated
Sponsor: Johnson & Johnson Consumer Inc. (J&JCI) (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CO-170302131230-URCT
Record Dates: First submitted 2017-11-08; First posted 2017-11-13 (Actual); Results first posted 2019-06-04 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-06

CONDITIONS: Common Cold
MeSH Terms: conditions — Common Cold

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- New Formulation Phenylephrine HCl (Experimental)
  Interventions: Drug: New Formulation Phenylephrine HCl
- Marketed Phenylephrine HCl (Active Comparator)
  Interventions: Drug: Marketed Phenylephrine HCl
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: New Formulation Phenylephrine HCl — 2 doses of one tablet 12 hours apart
  Arms: New Formulation Phenylephrine HCl
Drug: Marketed Phenylephrine HCl — 4 doses of one capsule 4 hours apart
  Arms: Marketed Phenylephrine HCl
Drug: Placebo — 4 doses of placebo capsule and tablet taken 4 hours apart
  Arms: Placebo

SUMMARY:
This will be a randomized, double-blind, placebo controlled, parallel-group Phase 2 study to evaluate the efficacy of a new formulation of phenylephrine HCl and a currently marketed phenylephrine HCl for relief of nasal congestion in subjects with naturally occurring cold symptoms.

ELIGIBILITY:
1. Provide a signed and dated informed consent form before any study-related procedures.
2. Men or non-pregnant, non-lactating women, aged 18 years or older, who have cold symptoms due to an acute upper respiratory tract infection but are otherwise healthy
3. Have experienced onset of common cold symptoms (per subject report) within 72 hours before study entry consisting of cold symptoms per the following:

   1. At Visit 1, at least moderate severity (score ≥ 5, on a scale from 0 = none to 7 = severe) for stuffy/congested nose, and
   2. At Visit 1, at least mild (score ≥ 3, on a scale from 0 = none to 7 = severe) for sinus pressure/tenderness, and
   3. Within the past 72 hours, two or more of the following symptoms: runny nose, sore or scratchy throat, sneezing, headache, malaise, or cough.
4. Are normotensive and have no clinically significant abnormalities identified by medical history or vital sign measurement (except as consistent with the diagnosis of the common cold) as determined by the Investigator at screening.

   * Blood pressure must be within the following limits after sitting for approximately 5 minutes: > 90 and <140 mm Hg systolic, and >50 and <90 mm Hg diastolic, at screening
   * Pulse rate >50 and <90 beats/minute at screening;
   * Body Mass Index (BMI) of 18 to 34 kg/m2 (inclusive);
5. Willing to use only the study treatment for cold symptom relief during the course of the study and avoid the use of treatments that may affect nasal / cold symptomatology; no other cough, cold, allergy, or analgesic/antipyretic medicines (non-prescription or prescription) or herbal/dietary supplements will be permitted during the study
6. Females of childbearing potential must have used an effective form of birth control for three months before Screening and a negative urine pregnancy test at the Screening visit.
7. Female and male subjects must agree to the contraceptive requirement use during the study and for at least 30 days after the last dose (for females) (See Section 10.4.3 ).
8. Willing and able to comply with the study procedures and visit schedule, which includes remaining at the study site for at least 4 hours after the first dose of study medicine on Day 1.
9. Able to read and understand English and/or French;

Exclusion criteria:

1. Currently experiencing nasal congestion due to allergic rhinitis or chronic respiratory disease.
2. Any ear, nose, throat, or respiratory tract disease, other than the common cold, identified by signs and symptoms reported by the subject, or by medical history or medication history
3. Presence of asthma.
4. History of rhinitis medicamentosa, anatomical nasal obstruction or deformity, nasal reconstructive surgery, or chronic sleep apnea.
5. Fever of ≥ 101.0 °F (38.3 °C).
6. Heart disease, controlled or uncontrolled hypertension, thyroid disease, diabetes, glaucoma, prostatic hypertrophy, or presence of a disease, which in the opinion of the investigator, would preclude the use of phenylephrine.
7. Are currently taking, or have taken within two weeks of screening, a monoamine oxidase inhibitor (MAOI).
8. Have the need to use medications which may impact nasal symptomatology i.e. systemic, inhaled (oral or nasal) corticosteroids, and the following drugs with significant anticholinergic properties: tricyclic antidepressants, paroxetine, medicines used to treat overactive bladder, antipsychotic medication, skeletal muscle relaxants, antiparkinsonian medication, the anticonvulsants carbamazepine and oxcarbazepine, and dicycloverine (dicyclomine), dimenhydrinate, propantheline, atropine, hyoscyamine, belladonna, prochlorperazine and promethazine.
9. Have a bacterial sinus infection within 2 weeks prior to screening.
10. Use of systemic antibiotics within the past 7 days prior to screening.
11. Known or suspected alcohol or substance abuse (e.g., amphetamines, benzodiazepines, cocaine, marijuana, opiates).
12. Use of marijuana containing substances within the 10 days prior to screening and throughout the study.
13. Positive Urine Drug Screen.
14. Use of alcohol throughout the study.
15. History of smoking tobacco products or use of nicotine-containing substances within the previous three months as determined by subject's medical history or subject's verbal report.
16. Known sensitivity to the investigational product or any excipients of the drug product.
17. Before the first dose of study medicine, use of

    1. oral or intranasal cold, cough, allergy, or analgesic/antipyretic medicines within approximately 12 hours;
    2. menthol products, medicated lozenge, humidifier, nasal saline spray or throat spray within approximately 6 hours;
    3. herbal/dietary supplements within approximately 12 hours.
18. Have difficulty swallowing tablets/capsules or are unable to swallow whole without crushing, chewing, splitting, or dissolving.
19. Subjects who were previously randomized and received the IP.
20. Significant unstable or uncontrolled medical condition that may interfere with a subject's participation in the study.
21. Other severe, acute or chronic, medical or psychiatric condition(s) or laboratory abnormality that may increase the risk associated with study participation or IP administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.
22. Currently participating in another clinical trial or has done so in the past 30 days.
23. Subjects who are related to those persons involved directly or indirectly with the conduct of this study (i.e., principal investigator, sub-investigators, study coordinators, other site personnel, employees of Johnson & Johnson (J&J) subsidiaries, contractors of J&J, and the families of each).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2017-11-30 (Actual); Primary Completion 2018-04-16 (Actual); Study Completion 2018-04-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steve Sacavage, Study Director — Johnson and Johnson Consumer, Inc
Locations (11):
- Canada (11):
  - The Medical Arts Health Research Group, Kelowna, British Columbia
  - Mission Hills Urgent Care Walk in Clinic, Mission, British Columbia
  - James Lai, MD, Inc, Vancouver, British Columbia
  - NEOMO Research, Greater Sudbury, Ontario
  - Dawson Road Family Medical Clinic, Guelph, Ontario
  - Sunningdale Health and Wellness Centre, London, Ontario
  - Bluewater Clinical Research Group, Inc., Sarnia, Ontario
  - Canadian Phase Onward, Inc., Toronto, Ontario
  - PrimeHealth Clinical Research, Toronto, Ontario
  - Diex Recherche, Sherbrooke, Quebec
  - Diex Recherche, Victoriaville, Quebec

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: One Placebo Extended-Release Tablet + One Placebo Immediate-Release Capsule Taken Orally Four Times Daily.
- PE-IR: One Phenylephrine HCl Immediate-Release Capsule + One Placebo Extended-Release Tablet Taken Orally Four Times Daily.
- PE-ER: One Phenylephrine HCl Extended-Release Tablet + One Placebo Immediate-Release Capsule Taken Orally Twice Daily AND One Placebo Extended-Release Tablet + One Placebo Immediate-Release Capsule Taken Orally Twice Daily.
Period: Overall Study
Arm/Group | Placebo | PE-IR | PE-ER
Started | 64 | 66 | 63
Completed | 63 | 65 | 63
Not Completed | 1 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | PE-IR | PE-ER | Total
Number analyzed (Participants) | 64 | 66 | 63 | 193
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.7 (14.60) | 43.4 (14.71) | 46.4 (15.44) | 44.8 (14.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 37 | 38 | 122
  Male | 17 | 29 | 25 | 71
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 2 | 3 | 10
  Not Hispanic or Latino | 59 | 64 | 60 | 183
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 3 | 1 | 6
  Asian | 7 | 11 | 7 | 25
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 3 | 0 | 5
  White | 50 | 48 | 53 | 151
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 1 | 2 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  North America: CAN | 64 | 66 | 63 | 193

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in the Nasal Congestion Severity Score
Description: Average change from baseline in the Nasal Congestion Severity Score on an 8 point scale with 0=None and 7=Severe. Change from baseline in the Nasal Congestion Severity Score averaged over assessments at 2, 4, 6, 8, 10, and 12 hours.
Time Frame: 0-12 hours
Population: Analysis is based on the Full Analysis Set population, which included all participants who were randomized and provided a valid baseline assessment of nasal congestion severity.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | PE-IR | PE-ER
Number analyzed (Participants) | 64 | 66 | 63
units on a scale | 1.80 (0.156) | 2.03 (0.154) | 1.93 (0.158)
Statistical Analysis 1: Comparison: Placebo vs PE-IR; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority; p = 0.300, ANOVA — The significance threshold level was 0.05 (two sided); Treatment and baseline nasal congestion score were factors; Mean Difference (Final Values) = 0.23, 95% CI 2-sided [-0.205 to 0.662], Standard Error of Mean 0.220
Statistical Analysis 2: Comparison: Placebo vs PE-ER; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority; p = 0.569, ANOVA — The significance threshold level was 0.05 (two sided); Treatment and baseline nasal congestion score were factors; Mean Difference (Final Values) = 0.13, 95% CI 2-sided [-0.311 to 0.564], Standard Error of Mean 0.222
Statistical Analysis 3: Comparison: PE-IR vs PE-ER; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority; p = 0.645, ANOVA — The significance threshold level was 0.05 (two sided); Treatment and baseline nasal congestion score were factors; Mean Difference (Final Values) = -0.10, 95% CI 2-sided [-0.537 to 0.333], Standard Error of Mean 0.220

2. Secondary Outcome: Average Change From Baseline in the Nasal Congestion Severity Score
Description: Average change from baseline in the Nasal Congestion Severity Score averaged over hours 8-12. This is an 8 point scale with 0=None and 7=Severe.
Time Frame: 0-12 hours
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | PE-IR | PE-ER
Number analyzed (Participants) | 64 | 66 | 63
units on a scale | 2.14 (0.185) | 2.39 (0.182) | 2.16 (0.187)
Statistical Analysis 1: Comparison: Placebo vs PE-IR; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority; p = 0.346, ANOVA — The significance threshold level was 0.05 (two sided); Treatment and baseline nasal congestion score were factors; Mean Difference (Final Values) = 0.25, 95% CI 2-sided [-0.267 to 0.759], Standard Error of Mean 0.260
Statistical Analysis 2: Comparison: Placebo vs PE-ER; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority; p = 0.938, ANOVA — The significance threshold level was 0.05 (two sided); Treatment and baseline nasal congestion score were factors; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-0.498 to 0.539], Standard Error of Mean 0.263
Statistical Analysis 3: Comparison: PE-IR vs PE-ER; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority; p = 0.389, ANOVA — The significance threshold level was 0.05 (two sided); Treatment and baseline nasal congestion score were factors; Mean Difference (Final Values) = -0.23, 95% CI 2-sided [-0.741 to 0.289], Standard Error of Mean 0.261

3. Secondary Outcome: Change From Baseline in the Nasal Congestion Severity Score
Description: Change from baseline in the Nasal Congestion Severity Score at 2 hours. This is an 8 point scale with 0=None and 7=Severe.
Time Frame: 0-2 hours
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | PE-IR | PE-ER
Number analyzed (Participants) | 64 | 66 | 63
units on a scale | 1.12 (0.163) | 1.24 (0.161) | 1.52 (0.165)
Statistical Analysis 1: Comparison: Placebo vs PE-IR; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority; p = 0.607, ANOVA; Treatment and baseline nasal congestion score were factors; Mean Difference (Final Values) = 0.12, 95% CI 2-sided [-0.33 to 0.57], Standard Error of Mean 0.230
Statistical Analysis 2: Comparison: Placebo vs PE-ER; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority; p = 0.085, ANOVA — The significance threshold level was 0.05 (two sided); Treatment and baseline nasal congestion score were factors; Mean Difference (Final Values) = 0.40, 95% CI 2-sided [-0.06 to 0.86], Standard Error of Mean 0.232
Statistical Analysis 3: Comparison: PE-IR vs PE-ER; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority; p = 0.220, ANOVA — The significance threshold level was 0.05 (two sided); Treatment and baseline nasal congestion score were factors; Mean Difference (Final Values) = 0.28, 95% CI 2-sided [-0.17 to 0.74], Standard Error of Mean 0.230

4. Secondary Outcome: Change From Baseline in the Nasal Congestion Severity Score
Description: Change from baseline in the Nasal Congestion Severity Score at 4 hours. This is an 8 point scale with 0=None and 7=Severe.
Time Frame: 0-4 hours
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | PE-IR | PE-ER
Number analyzed (Participants) | 64 | 66 | 63
units on a scale | 1.69 (0.193) | 1.82 (0.190) | 1.71 (0.194)
Statistical Analysis 1: Comparison: Placebo vs PE-IR; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority; p = 0.633, ANOVA — The significance threshold level was 0.05 (two sided); Treatment and baseline nasal congestion score were factors; Mean Difference (Final Values) = 0.13, 95% CI 2-sided [-0.40 to 0.66], Standard Error of Mean 0.271
Statistical Analysis 2: Comparison: Placebo vs PE-ER; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority; p = 0.952, ANOVA — The significance threshold level was 0.05 (two sided); Treatment and baseline nasal congestion score were factors; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-0.52 to 0.56], Standard Error of Mean 0.273
Statistical Analysis 3: Comparison: PE-IR vs PE-ER; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority; p = 0.678, ANOVA — The significance threshold level was 0.05 (two sided); Treatment and baseline nasal congestion score were factors; Mean Difference (Final Values) = -0.11, 95% CI 2-sided [-0.65 to 0.42], Standard Error of Mean 0.272

5. Secondary Outcome: Change From Baseline in the Nasal Congestion Severity Score
Description: Change from baseline in the Nasal Congestion Severity Score at 6 hours. This is an 8 point scale with 0=None and 7=Severe.
Time Frame: 0-6 hours
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | PE-IR | PE-ER
Number analyzed (Participants) | 64 | 66 | 63
units on a scale | 1.58 (0.178) | 1.97 (0.176) | 1.86 (0.180)
Statistical Analysis 1: Comparison: Placebo vs PE-IR; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority; p = 0.126, ANOVA — The significance threshold level was 0.05 (two sided); Treatment and baseline nasal congestion score were factors; Mean Difference (Final Values) = 0.38, 95% CI 2-sided [-0.11 to 0.88], Standard Error of Mean 0.250
Statistical Analysis 2: Comparison: Placebo vs PE-ER; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority; p = 0.270, ANOVA — The significance threshold level was 0.05 (two sided); Treatment and baseline nasal congestion score were factors; Mean Difference (Final Values) = 0.28, 95% CI 2-sided [-0.22 to 0.78], Standard Error of Mean 0.253
Statistical Analysis 3: Comparison: PE-IR vs PE-ER; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority; p = 0.676, ANOVA — The significance threshold level was 0.05 (two sided); Treatment and baseline nasal congestion score were factors; Mean Difference (Final Values) = -0.11, 95% CI 2-sided [-0.60 to 0.39], Standard Error of Mean 0.251

6. Secondary Outcome: Change From Baseline in the Nasal Congestion Severity Score
Description: Change from baseline in the Nasal Congestion Severity Score at 8 hours. This is an 8 point scale with 0=None and 7=Severe.
Time Frame: 0-8 hours
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | PE-IR | PE-ER
Number analyzed (Participants) | 64 | 66 | 63
units on a scale | 2.00 (0.188) | 2.22 (0.185) | 1.99 (0.189)
Statistical Analysis 1: Comparison: Placebo vs PE-IR; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority; p = 0.421, ANOVA — The significance threshold level was 0.05 (two sided); Treatment and baseline nasal congestion score were factors; Mean Difference (Final Values) = 0.21, 95% CI 2-sided [-0.31 to 0.73], Standard Error of Mean 0.264
Statistical Analysis 2: Comparison: Placebo vs PE-ER; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority; p = 0.970, ANOVA — The significance threshold level was 0.05 (two sided); Treatment and baseline nasal congestion score were factors; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.54 to 0.52], Standard Error of Mean 0.266
Statistical Analysis 3: Comparison: PE-IR vs PE-ER; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority; p = 0.401, ANOVA — The significance threshold level was 0.05 (two sided); Treatment and baseline nasal congestion score were factors; Mean Difference (Final Values) = -0.22, 95% CI 2-sided [-0.74 to 0.30], Standard Error of Mean 0.265

7. Secondary Outcome: Change From Baseline in the Nasal Congestion Severity Score
Description: Change from baseline in the Nasal Congestion Severity Score at 10 hours. This is an 8 point scale with 0=None and 7=Severe.
Time Frame: 0-10 hours
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | PE-IR | PE-ER
Number analyzed (Participants) | 64 | 66 | 63
units on a scale | 2.14 (0.193) | 2.45 (0.191) | 2.18 (0.195)
Statistical Analysis 1: Comparison: Placebo vs PE-IR; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority; p = 0.257, ANOVA — The significance threshold level was 0.05 (two sided); Treatment and baseline nasal congestion score were factors; Mean Difference (Final Values) = 0.31, 95% CI 2-sided [-0.23 to 0.85], Standard Error of Mean 0.272
Statistical Analysis 2: Comparison: Placebo vs PE-ER; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority; p = 0.877, ANOVA — The significance threshold level was 0.05 (two sided); Treatment and baseline nasal congestion score were factors; Mean Difference (Final Values) = 0.04, 95% CI 2-sided [-0.50 to 0.58], Standard Error of Mean 0.275
Statistical Analysis 3: Comparison: PE-IR vs PE-ER; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority; p = 0.329, ANOVA — The significance threshold level was 0.05 (two sided); Treatment and baseline nasal congestion score were factors; Mean Difference (Final Values) = -0.27, 95% CI 2-sided [-0.80 to 0.27], Standard Error of Mean 0.273

8. Secondary Outcome: Change From Baseline in the Nasal Congestion Severity Score
Description: Change from baseline in the Nasal Congestion Severity Score at 12 hours. This is an 8 point scale with 0=None and 7=Severe.
Time Frame: 0-12 hours
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | PE-IR | PE-ER
Number analyzed (Participants) | 64 | 66 | 63
units on a scale | 2.28 (0.212) | 2.50 (0.209) | 2.31 (0.214)
Statistical Analysis 1: Comparison: Placebo vs PE-IR; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority; p = 0.469, ANOVA — The significance threshold level was 0.05 (two sided); Treatment and baseline nasal congestion score were factors; Mean Difference (Final Values) = 0.22, 95% CI 2-sided [-0.37 to 0.80], Standard Error of Mean 0.298
Statistical Analysis 2: Comparison: Placebo vs PE-ER; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority; p = 0.924, ANOVA — The significance threshold level was 0.05 (two sided); Treatment and baseline nasal congestion score were factors; Mean Difference (Final Values) = 0.03, 95% CI 2-sided [-0.57 to 0.62], Standard Error of Mean 0.301
Statistical Analysis 3: Comparison: PE-IR vs PE-ER; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority; p = 0.532, ANOVA — The significance threshold level was 0.05 (two sided); Treatment and baseline nasal congestion score were factors; Mean Difference (Final Values) = -0.19, 95% CI 2-sided [-0.78 to 0.40], Standard Error of Mean 0.299

9. Secondary Outcome: Change From Baseline in the Nasal Congestion Severity Score
Description: Change from baseline in the Nasal Congestion Severity Score at 24 hours. This is an 8 point scale with 0=None and 7=Severe.
Time Frame: 0-24 hours
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | PE-IR | PE-ER
Number analyzed (Participants) | 64 | 66 | 63
units on a scale | 2.78 (0.220) | 2.61 (0.217) | 2.52 (0.222)
Statistical Analysis 1: Comparison: Placebo vs PE-IR; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority; p = 0.579, ANOVA — The significance threshold level was 0.05 (two sided); Treatment and baseline nasal congestion score were factors; Mean Difference (Final Values) = -0.17, 95% CI 2-sided [-0.78 to 0.44], Standard Error of Mean 0.309
Statistical Analysis 2: Comparison: Placebo vs PE-ER; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority; p = 0.394, ANOVA — The significance threshold level was 0.05 (two sided); Treatment and baseline nasal congestion score were factors; Mean Difference (Final Values) = -0.27, 95% CI 2-sided [-0.88 to 0.35], Standard Error of Mean 0.312
Statistical Analysis 3: Comparison: PE-IR vs PE-ER; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority; p = 0.760, ANOVA — The significance threshold level was 0.05 (two sided); Treatment and baseline nasal congestion score were factors; Mean Difference (Final Values) = -0.09, 95% CI 2-sided [-0.71 to 0.52], Standard Error of Mean 0.310

10. Secondary Outcome: Average Change From Baseline in Sinus Pressure/Tenderness Scores
Description: Change from baseline in Sinus Pressure/Tenderness Scores averaged over assessments at 2, 4, 6, 8, 10, and 12 hours. This is an 8 point scale with 0=None and 7=Severe.
Time Frame: 0-12 hours
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | PE-IR | PE-ER
Number analyzed (Participants) | 64 | 66 | 63
units on a scale | 1.67 (0.155) | 1.78 (0.152) | 1.74 (0.156)
Statistical Analysis 1: Comparison: Placebo vs PE-IR; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority; p = 0.616, ANCOVA — The significance threshold level was 0.05 (two sided); Treatment and baseline sinus pressure/tenderness score were factors; Mean Difference (Final Values) = 0.11, 95% CI 2-sided [-0.320 to 0.539], Standard Error of Mean 0.218
Statistical Analysis 2: Comparison: Placebo vs PE-ER; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority; p = 0.734, ANCOVA — The significance threshold level was 0.05 (two sided); Treatment and baseline sinus pressure/tenderness score were factors; Mean Difference (Final Values) = 0.07, 95% CI 2-sided [-0.359 to 0.508], Standard Error of Mean 0.220
Statistical Analysis 3: Comparison: PE-IR vs PE-ER; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority; p = 0.874, ANCOVA — The significance threshold level was 0.05 (two sided); Treatment and baseline sinus pressure/tenderness score were factors; Mean Difference (Final Values) = -0.03, 95% CI 2-sided [-0.465 to 0.395], Standard Error of Mean 0.218

11. Secondary Outcome: Change From Baseline in Sinus Pressure/Tenderness Scores
Description: Change from baseline in Sinus Pressure/Tenderness Scores at 2 hours. This is an 8 point scale with 0=None and 7=Severe.
Time Frame: 0-2 hours
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | PE-IR | PE-ER
Number analyzed (Participants) | 64 | 66 | 63
units on a scale | 1.10 (0.163) | 1.03 (0.161) | 1.30 (0.164)
Statistical Analysis 1: Comparison: Placebo vs PE-IR; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority; p = 0.750, ANCOVA — The significance threshold level was 0.05 (two sided); Treatment and baseline sinus pressure/tenderness score were factors; Mean Difference (Final Values) = -0.07, 95% CI 2-sided [-0.53 to 0.38], Standard Error of Mean 0.230
Statistical Analysis 2: Comparison: Placebo vs PE-ER; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority; p = 0.390, ANCOVA — The significance threshold level was 0.05 (two sided); Treatment and baseline sinus pressure/tenderness score were factors; Mean Difference (Final Values) = 0.20, 95% CI 2-sided [-0.26 to 0.66], Standard Error of Mean 0.232
Statistical Analysis 3: Comparison: PE-IR vs PE-ER; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority; p = 0.236, ANCOVA — The significance threshold level was 0.05 (two sided); Treatment and baseline sinus pressure/tenderness score were factors; Mean Difference (Final Values) = 0.27, 95% CI 2-sided [-0.18 to 0.73], Standard Error of Mean 0.230

12. Secondary Outcome: Change From Baseline in Sinus Pressure/Tenderness Scores
Description: Change from baseline in Sinus Pressure/Tenderness Scores at 4 hours.
Time Frame: 0-4 hours
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | PE-IR | PE-ER
Number analyzed (Participants) | 64 | 66 | 63
units on a scale | 1.54 (0.190) | 1.43 (0.187) | 1.48 (0.191)
Statistical Analysis 1: Comparison: Placebo vs PE-IR; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority; p = 0.707, ANCOVA — The significance threshold level was 0.05 (two sided); Treatment and baseline sinus pressure/tenderness score were factors; Mean Difference (Final Values) = -0.10, 95% CI 2-sided [-0.63 to 0.43], Standard Error of Mean 0.267
Statistical Analysis 2: Comparison: Placebo vs PE-ER; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority; p = 0.839, ANCOVA — The significance threshold level was 0.05 (two sided); Treatment and baseline sinus pressure/tenderness score were factors; Mean Difference (Final Values) = -0.05, 95% CI 2-sided [-0.59 to 0.48], Standard Error of Mean 0.269
Statistical Analysis 3: Comparison: PE-IR vs PE-ER; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority; p = 0.864, ANCOVA — The significance threshold level was 0.05 (two sided); Treatment and baseline sinus pressure/tenderness score were factors; Mean Difference (Final Values) = 0.05, 95% CI 2-sided [-0.48 to 0.57], Standard Error of Mean 0.267

13. Secondary Outcome: Change From Baseline in Sinus Pressure/Tenderness Scores
Description: Change from baseline in Sinus Pressure/Tenderness Scores at 6 hours. This is an 8 point scale with 0=None and 7=Severe.
Time Frame: 0-6 hours
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | PE-IR | PE-ER
Number analyzed (Participants) | 64 | 66 | 63
units on a scale | 1.62 (0.181) | 1.69 (0.179) | 1.75 (0.182)
Statistical Analysis 1: Comparison: Placebo vs PE-IR; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority; p = 0.794, ANCOVA — The significance threshold level was 0.05 (two sided); Treatment and baseline sinus pressure/tenderness score were factors; Mean Difference (Final Values) = 0.07, 95% CI 2-sided [-0.44 to 0.57], Standard Error of Mean 0.255
Statistical Analysis 2: Comparison: Placebo vs PE-ER; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority; p = 0.628, ANCOVA — The significance threshold level was 0.05 (two sided); Treatment and baseline sinus pressure/tenderness score were factors; Mean Difference (Final Values) = 0.12, 95% CI 2-sided [-0.38 to 0.63], Standard Error of Mean 0.257
Statistical Analysis 3: Comparison: PE-IR vs PE-ER; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority; p = 0.820, ANCOVA — The significance threshold level was 0.05 (two sided); Treatment and baseline sinus pressure/tenderness score were factors; Mean Difference (Final Values) = 0.06, 95% CI 2-sided [-0.45 to 0.56], Standard Error of Mean 0.255

14. Secondary Outcome: Change From Baseline in Sinus Pressure/Tenderness Scores
Description: Change from baseline in Sinus Pressure/Tenderness Scores at 8 hours. This is an 8 point scale with 0=None and 7=Severe.
Time Frame: 0-8 hours
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | PE-IR | PE-ER
Number analyzed (Participants) | 64 | 66 | 63
units on a scale | 1.69 (0.189) | 1.95 (0.186) | 1.82 (0.190)
Statistical Analysis 1: Comparison: Placebo vs PE-IR; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority; p = 0.330, ANCOVA — The significance threshold level was 0.05 (two sided); Treatment and baseline sinus pressure/tenderness score were factors; Mean Difference (Final Values) = 0.26, 95% CI 2-sided [-0.27 to 0.79], Standard Error of Mean 0.266
Statistical Analysis 2: Comparison: Placebo vs PE-ER; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority; p = 0.631, ANCOVA — The significance threshold level was 0.05 (two sided); Treatment and baseline sinus pressure/tenderness score were factors; Mean Difference (Final Values) = 0.13, 95% CI 2-sided [-0.40 to 0.66], Standard Error of Mean 0.269
Statistical Analysis 3: Comparison: PE-IR vs PE-ER; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority; p = 0.625, ANCOVA — The significance threshold level was 0.05 (two sided); Treatment and baseline sinus pressure/tenderness score were factors; Mean Difference (Final Values) = -0.13, 95% CI 2-sided [-0.66 to 0.40], Standard Error of Mean 0.266

15. Secondary Outcome: Change From Baseline in Sinus Pressure/Tenderness Scores
Description: Change from baseline in Sinus Pressure/Tenderness Scores at 10 hours. This is an 8 point scale with 0=None and 7=Severe.
Time Frame: 0-10 hours
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on scale
Arm/Group | Placebo | PE-IR | PE-ER
Number analyzed (Participants) | 64 | 66 | 63
units on scale | 1.91 (0.196) | 2.23 (0.193) | 1.96 (0.197)
Statistical Analysis 1: Comparison: Placebo vs PE-IR; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority; p = 0.240, ANCOVA — The significance threshold level was 0.05 (two sided); Treatment and baseline sinus pressure/tenderness score were factors; Mean Difference (Final Values) = 0.32, 95% CI 2-sided [-0.22 to 0.87], Standard Error of Mean 0.275
Statistical Analysis 2: Comparison: Placebo vs PE-IR; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority; p = 0.865, ANCOVA — The significance threshold level was 0.05 (two sided); Treatment and baseline sinus pressure/tenderness score were factors; Mean Difference (Final Values) = 0.05, 95% CI 2-sided [-0.50 to 0.60], Standard Error of Mean 0.278
Statistical Analysis 3: Comparison: PE-IR vs PE-ER; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority; p = 0.316, ANCOVA — The significance threshold level was 0.05 (two sided); Treatment and baseline sinus pressure/tenderness score were factors; Mean Difference (Final Values) = -0.28, 95% CI 2-sided [-0.82 to 0.27], Standard Error of Mean 0.275

16. Secondary Outcome: Change From Baseline in Sinus Pressure/Tenderness Scores
Description: Change from baseline in Sinus Pressure/Tenderness Scores at 12 hours. This is an 8 point scale with 0=None and 7=Severe.
Time Frame: 0-12 hours
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | PE-IR | PE-ER
Number analyzed (Participants) | 64 | 66 | 63
units on a scale | 2.15 (0.202) | 2.32 (0.199) | 2.15 (0.203)
Statistical Analysis 1: Comparison: Placebo vs PE-IR; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority; p = 0.529, ANCOVA — The significance threshold level was 0.05 (two sided); Treatment and baseline sinus pressure/tenderness score were factors; Mean Difference (Final Values) = 0.18, 95% CI 2-sided [-0.38 to 0.74], Standard Error of Mean 0.284
Statistical Analysis 2: Comparison: Placebo vs PE-ER; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority; p = 0.997, ANCOVA — The significance threshold level was 0.05 (two sided); Treatment and baseline sinus pressure/tenderness score were factors; Mean Difference (Final Values) = 0.00, 95% CI 2-sided [-0.56 to 0.57], Standard Error of Mean 0.287
Statistical Analysis 3: Comparison: PE-IR vs PE-ER; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority; p = 0.532, ANCOVA — The significance threshold level was 0.05 (two sided); Treatment and baseline sinus pressure/tenderness score were factors; Mean Difference (Final Values) = -0.18, 95% CI 2-sided [-0.74 to 0.38], Standard Error of Mean 0.285

17. Secondary Outcome: Change From Baseline in Sinus Pressure/Tenderness Scores
Description: Change from baseline in Sinus Pressure/Tenderness Scores at 24 hours. This is an 8 point scale with 0=None and 7=Severe.
Time Frame: 0-24 hours
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | PE-IR | PE-ER
Number analyzed (Participants) | 64 | 66 | 63
units on a scale | 2.61 (0.220) | 2.39 (0.216) | 2.23 (0.221)
Statistical Analysis 1: Comparison: Placebo vs PE-IR; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority; p = 0.468, ANCOVA — The significance threshold level was 0.05 (two sided); Treatment and baseline sinus pressure/tenderness score were factors; Mean Difference (Final Values) = -0.22, 95% CI 2-sided [-0.83 to 0.38], Standard Error of Mean 0.309
Statistical Analysis 2: Comparison: Placebo vs PE-ER; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority; p = 0.218, ANCOVA — The significance threshold level was 0.05 (two sided); Treatment and baseline sinus pressure/tenderness score were factors; Mean Difference (Final Values) = -0.39, 95% CI 2-sided [-1.00 to 0.23], Standard Error of Mean 0.312
Statistical Analysis 3: Comparison: PE-IR vs PE-ER; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority; p = 0.604, ANCOVA — The significance threshold level was 0.05 (two sided); Treatment and baseline sinus pressure/tenderness score were factors; Mean Difference (Final Values) = -0.16, 95% CI 2-sided [-0.77 to 0.45], Standard Error of Mean 0.309

ADVERSE EVENTS:
Time Frame: Within three days for nonserious adverse events, +30 days after the participant's last dose or exposure to the investigational product for serious adverse events.
Description: AEs were systematically collected during the study and at the follow-up visit at Day 2 (+/-1 day). Spontaneously reported AEs collected during the study were also recorded. Any clinically important abnormalities or causally-related AEs persisting were followed until resolution or until reaching a clinically stable endpoint.
Arm/Group | Placebo | PE-IR | PE-ER
All-Cause Mortality (participants affected / at risk) | 0/64 | 0/66 | 0/63
Serious Adverse Events (participants affected / at risk) | 0/64 | 0/66 | 0/63
Other Adverse Events (participants affected / at risk) | 0/64 | 0/66 | 0/63

LIMITATIONS AND CAVEATS:
An interim statistical analysis was conducted after the study failed to meet planned enrollment in the 2017-2018 cold season. The study was subsequently cancelled and enrollment was discontinued. Analysis of the 193 enrolled subjects was conducted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2018-06-14): https://cdn.clinicaltrials.gov/large-docs/26/NCT03339726/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-31): https://cdn.clinicaltrials.gov/large-docs/26/NCT03339726/SAP_001.pdf